CLINICAL TRIAL: NCT07303660
Title: A Phase 1b Study of Lonitoclax + Azacitidine (Aza) in Acute Myeloid Leukemia (AML) Patients
Brief Title: A Phase 1b Study of Lonitoclax + Azacitidine in Acute Myeloid Leukemia Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lomond Therapeutics Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZE50-0134-0004
Record Dates: First submitted 2025-12-05; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose optimization study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- ZE50-0134 + Azacitidine Dose Level -1 (Experimental): Optional and would only be performed Dose Level 1 is poorly tolerated.
  Interventions: Drug: Azacitidine Days 1-7; Drug: ZE 50-0134
- ZE50-0134 + Azacitidine Dose Level 1 (Experimental)
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7
- ZE50-0134 + Azacitidine Dose Level 2 (Experimental)
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7
- ZE50-0134 + Azacitidine Dose Level 3 (Experimental)
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7
- ZE50-0134 + Azacitidine Dose Level 4 (Experimental)
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7
- ZE50-0134 + Azacitidine Dose Level 5 (Experimental)
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7
- ZE50-0134 + Azacitidine Selected dose 1 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study.
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7
- ZE50-0134 + Azacitidine Selected dose 2 (Experimental): The doses used in Part 2 of the study will be determined based on the data from Part 1 of the study.
  Interventions: Drug: ZE50-0134; Drug: Azacitidine Days 1-7

INTERVENTIONS:
Drug: ZE50-0134 — Oral capsules BID
  Arms: ZE50-0134 + Azacitidine Dose Level 1; ZE50-0134 + Azacitidine Dose Level 2; ZE50-0134 + Azacitidine Dose Level 3; ZE50-0134 + Azacitidine Dose Level 4; ZE50-0134 + Azacitidine Dose Level 5; ZE50-0134 + Azacitidine Selected dose 1; ZE50-0134 + Azacitidine Selected dose 2
Drug: Azacitidine Days 1-7 — 75 mg/m2 daily, days 1-7
Drug: ZE 50-0134 — Oral capsules QD
  Arms: ZE50-0134 + Azacitidine Dose Level -1

SUMMARY:
This is a clinical study aiming to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of ZE50-0134 in relapsed and refractory Acute Myeloid Leukemia patients.

DETAILED DESCRIPTION:
It is an open-label Phase 1b clinical study of Lonitoclax + Aza in relapsed/refractory AML patients. The study is an open-label, with 2 parts.

The phase 1b dose escalation portion would include relapsed/refractory patients, as well as in the expansion group. Once the phase 1b dose and schedule of Lonitoclax + Aza is defined in the 3 + 3 design with biologically effective dose assessment, an amendment will be filed with the Regulatory Authorities and expansion cohort of 30 relapsed and refractory AML patients would be enrolled at two different doses (15 patients per dose) to determine the RP2D; the first dosing will be at the presumed potential phase 2 dose combination and the second dosing will be below this.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand and provide written informed consent. 2. AML patients: For the dose escalation and expansion, patients aged 18 and older with relapsed and/or refractory AML would be eligible. Prior treatment with a hypomethylating agent or Venetoclax is allowed.

3. At the time of Lonitoclax initiation, white blood count (WBC) needs to be < 25 × 109/L: Hydroxyurea can be used to achieve that level.

4. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2. 5. Adequate organ function as defined by the following:

1. Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 2.5 x ULN. AST and/or ALT may be up to 5 x ULN if thought to be secondary to leukemia.
2. Total bilirubin ≤ 1.5 x ULN (patients with known Gilbert's syndrome may enroll if direct bilirubin is ≤ 3 x ULN) for the local laboratory.
3. Estimated Glomerular Filtration Rate (eGFR) according to the Chronic Kidney Disease Epidemiology Collaboration (CDK-EPI) ≥ 60 mL/min/1.73m2 for the local laboratory.

   6. Female patients of childbearing potential must agree to use a highly effective method of contraception from screening visit until 120 days following the last dose of study treatment. Highly effective methods of contraception include sexual abstinence, bilateral tubal ligation, tricycle combined (estrogen and progestogen containing) oral or transdermal hormonal contraceptives, intrauterine devices and vasectomized partner. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

   7. Male patients capable of having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use highly effective contraception from the screening visit until 120 days until the last dose of study treatment, and themselves use barrier contraception (i.e., condoms). They must also refrain from sperm donation from the screening visit until 120 days following the last dose of study treatment. Should his partner become pregnant or suspect she is pregnant while he is participating in this study, he should inform his treating physician immediately.

   8. Patients must be able to take oral medications. Exclusion Criteria
   1. Isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement with AML).
   2. Acute promyelocytic leukemia (FAB M3).
   3. Active central nervous system (CNS) involvement by AML.
   4. Clinical signs/symptoms of leukostasis requiring urgent therapy.
   5. Known active infection with Human Immunodeficiency Virus (HIV), hepatitis B or hepatitis C. Patients with a history of positive serology for hepatitis B or C require a negative Polymerase chain reaction (PCR) test for virus to go onto therapy.
   6. Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis
   7. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent; if the half-life of the agent is unknown, patients must wait 1 week prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by Regulatory Authorities.
   8. Systemic antineoplastic therapy within 1 week (or 5 half-lives of drug received, whichever is shorter) or radiation therapy within 1 week prior to starting protocol except for hydroxyurea, which is allowed to control white blood cell counts.
   9. Female patients who are pregnant or lactating.
   10. Patients with psychological, familial, social, or geographic factors, other significant medical condition, laboratory abnormality that otherwise preclude them from giving informed consent, following the protocol, potentially hamper compliance with study treatment and follow-up or would confound the interpretation of the results of the trial.
   11. Concomitant medications that are strong CYP3A4 inducers.
   12. Patients with QTcF > 470 msec that cannot be corrected with electrolyte replacement, hydration, or medication modifications. This does not apply to patients with a pacemaker as measurement of QTc is not accurate under such conditions and bears no risk to patients since they are being medically paced by their device.
   13. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction with evidence of residual abnormalities within 6 months prior to enrollment (Troponin leak alone not included if no residual dysfunction), familial QT prolongation, known potassium wasting syndrome (Bartter syndrome, Gitelman syndrome, and Liddle syndrome), New York Heart Association (NYHA) Class III or IV heart failure, electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
   14. As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.

   Exclusion Criteria:
   1. Isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement with AML).
   2. Acute promyelocytic leukemia (FAB M3).
   3. Active central nervous system (CNS) involvement by AML.
   4. Clinical signs/symptoms of leukostasis requiring urgent therapy.
   5. Known active infection with Human Immunodeficiency Virus (HIV), hepatitis B or hepatitis C. Patients with a history of positive serology for hepatitis B or C require a negative Polymerase chain reaction (PCR) test for virus to go onto therapy.
   6. Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis
   7. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent; if the half-life of the agent is unknown, patients must wait 1 week prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by Regulatory Authorities.
   8. Systemic antineoplastic therapy within 1 week (or 5 half-lives of drug received, whichever is shorter) or radiation therapy within 1 week prior to starting protocol except for hydroxyurea, which is allowed to control white blood cell counts.
   9. Female patients who are pregnant or lactating.
   10. Patients with psychological, familial, social, or geographic factors, other significant medical condition, laboratory abnormality that otherwise preclude them from giving informed consent, following the protocol, potentially hamper compliance with study treatment and follow-up or would confound the interpretation of the results of the trial.
   11. Concomitant medications that are strong CYP3A4 inducers.
   12. Patients with QTcF > 470 msec that cannot be corrected with electrolyte replacement, hydration, or medication modifications. This does not apply to patients with a pacemaker as measurement of QTc is not accurate under such conditions and bears no risk to patients since they are being medically paced by their device.
   13. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction with evidence of residual abnormalities within 6 months prior to enrollment (Troponin leak alone not included if no residual dysfunction), familial QT prolongation, known potassium wasting syndrome (Bartter syndrome, Gitelman syndrome, and Liddle syndrome), New York Heart Association (NYHA) Class III or IV heart failure, electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
   14. As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Determination of the RP2D and expansion cohort enrollment | Up to 24 cycles, 4 weeks each
  To determine the recommended phase 2 (RP2D) dose using a 28-day schedule in relapsed and refractory (R/R) AML followed by an expansion cohort.

SECONDARY OUTCOMES:
Composite response rate | Up to 24 cycles, 4 weeks each
  Composite response rate will be defined as the proportion of efficacy-evaluable patients who achieve CR, CRi, CRh, or MLFS.
To determine the time to neutrophil and platelet recovery in patients receiving Lonitoclax + Aza | Up to 24 cycles, 4 weeks each
  Monitoring of neutrophil and platelet counts
Overall incidence of treatment-related and non-treatment-related toxicities | Up to 24 cycles, 4 weeks each
  To determine the overall incidence of treatment-related and non-treatment-related toxicities.
Event-free survival | Up to 24 cycles, 4 weeks each
  Event-free survival will be measured from start of the treatment to the first of failure to achieve a CR/CRi/CRh/MLFS, or relapse, or death due to any cause, with patients last known to be alive and event-free censored at the date of last contact.
Duration of remission | Up to 24 cycles, 4 weeks each
  Duration of remission is defined in responders as the time from documentation of remission to the date of disease progression.

OTHER OUTCOMES:
The percentage of patients that undergo hematopoietic stem cell transplant (HSCT) | Up to 24 cycles, 4 weeks each
  To determine the percentage of patients that undergo hematopoietic stem cell transplant (HSCT).
Peak plasma concentration of Lonitoclax | 3 cycles, 4 weeks each
  To determine peak plasma concentration of Lonitoclax when dosed in combination with Aza and its interaction with strong CYP3A4 inhibitors used in this disease
Investigating the baseline properties of leukemia cells | Up to 24 cycles, 4 weeks each
  To examine the baseline properties of leukemia cells that respond versus those that do not respond to initial therapy.
Serial properties of AML cells | Up to 24 cycles, 4 weeks each
  To determine the serial properties of AML cells that respond and then become resistant to this novel combination.
Minimal Residual Disease (MRD) and immune effects | 3 and 6 cycles, 4 weeks each
  A BM aspirate and biopsy will be performed at time of count recovery or day 42 (whichever occurs first) after 3 and 6 total cycles of therapy (induction + continuation therapy cycles) and for MRD assessment done by a central lab.
Time to maximum concentration of Lonitoclax | 3 cycles, 4 weeks each
  To determin time to maximum concentration of Lonitoclax when dosed in combination with Aza and its interaction with strong CYP3A4 inhibitors used in this disease
Area Under the Curve | 3 cycles, 4 weeks each
  To determine Area Under the Curve of Lonitoclax when dosed in combination with Aza and its interaction with strong CYP3A4 inhibitors used in this disease
The half-life of Lonitoclax | 3 cycles, 4 weeks each
  To determine the half-life of Lonitoclax when dosed in combination with Aza and its interaction with strong CYP3A4 inhibitors used in this disease

IPD SHARING:
Plan to Share IPD: No